CLINICAL TRIAL: NCT07052110
Title: Listening to the Patient's Cancer Journey: A Randomised Controlled Trial of Digital Storytelling (DST) in Reducing Depressive Symptoms, Enhancing Self-esteem, and Promoting Quality of Life Among Hong Kong Chinese Childhood Cancer Survivors
Brief Title: A RCT of DST in Reducing Depressive Symptoms, Enhancing Self-esteem, and Promoting Quality of Life Among CCSs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hong Kong Children's Hospital (Other); Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DST intervention
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Cancer
Keywords: childhood cancer survivors; digitial storytelling; depressive symptoms; self-esteem; quality of life
MeSH Terms: conditions — Neoplasms; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Intervention Arm (Experimental): Participants in the experimental group will receive the DST intervention, which comprises four workshops. Each workshop will last 2.5 hours and will be conducted by a qualified interventionist. In the workshops, a group of 6-8 participants will first share their personal cancer experiences and offer feedback to other participants in the context of a story circle. A set of guiding questions will be used to facilitate participants in telling their own stories. Particularly, probing will be used to guide the child participants to share their own experiences. Open-ended questions such as 'How do you think about your cancer experience?' will be asked. Subsequent supplementary questions, such as 'What makes you feel in this way?' and 'can you give me some examples' will be asked to encourage more sharing. Afterwards, participants wil be encouraged to write their own script and storyboard, record their stories using a microphone, and choose photos and videos to illustrate their stories.
  Interventions: Other: Digital storytelling
- No Intervention: Control Arm (No Intervention): No intervention will be carried out among participants in the control group. However, customary care including medical follow-up, medication prescription, and nursing interventions will be provided, as usual.

INTERVENTIONS:
Other: Digital storytelling — DST is an intervention that can potentially mitigate the psychological impact of traumatic experiences. People can usually find positive meaning in a traumatic experience by communicating their experience using narratives like storytelling. In particular, by externalising the traumatic experience in the form of a narrative, the individual can become an objective agent, distancing themselves from negative meanings attached to the experience. This lowers people's resistance to and defence against the experience, assisting them to explore alternative perspectives regarding the experience and to identify its positive aspects, which boost self-esteem. Likewise, storytelling engages different areas of the brain, including those responsible for visual, language, and hearing functions, to reorganise the disorganised traumatic experience into a coherent story, facilitating integration of the experience into existing memories.
  Arms: Intervention: Intervention Arm

SUMMARY:
This study aims to examine the effectiveness of Digital storytelling (DST) in reducing depressive symptoms, enhancing self-esteem, and promoting quality of life among Chinese survivors of childhood cancer.

Participants in the experimental group will be divided into groups of 6 to 8 childhood cancer survivors to receive the intervention, which comprises four workshops. Each workshop will last 2.5 hours and will be conducted by a qualified interventionist. Parents are not required to attend the workshop. We will provide a waiting room for them. Parents will also be provided with a leaflet developed by Hong Kong Department of Health which contains self-help material for depression.

No intervention will be carried out among participants in the control group. However, customary care including medical follow-up, medication prescription, and nursing interventions will be provided, as usual. Parents will also be provided with a leaflet containing self-help materials for depression.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 13 and 18 years;
* (2) able to speak Cantonese and read Chinese; and
* (3) completed the active treatment of cancer.

Exclusion Criteria:

* survivors with mental and behavioural problems documented in their medical records.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms: Chinese version of the Center for Epidemiological Studies Depression Scale for Children (CES-DC) | The CES-DC will be conducted immediately after the completion of the intervention, and at 1-, 3- and 6-month follow-up via telephone interview.
  The CES-DC will be used to assess the number of depressive symptoms among participants. This instrument contains 20 items evaluated on a 4-point scale, from 0 (not at all) to 3 (a lot). The possible range of scores is between 0 and 60, with higher scores indicating more depressive symptoms. The cut-off score is 15. Participants with scores higher than 15 are considered to be experiencing significant levels of depressive symptoms. This scale has been widely applied in studies among Hong Kong Chinese children with cancer, and its psychometric properties have been well-established in this population.

SECONDARY OUTCOMES:
Self-esteem: Chinese version of the Rosenberg Self-Esteem Scale (RSES) | The RSES will be conducted immediately after the completion of the intervention, and at 1-, 3- and 6-month follow-up via telephone interview.
  The RSES will be used to assess participants' self-esteem. This scale contains 10 items that are evaluated on a scale of 1 to 4. Higher scores indicate higher levels of self-esteem. This scale has been widely applied in paediatric oncology research and has been previously validated in Hong Kong Chinese children.
Quality of life: Chinese version of the Pediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0) | The PedsQL 4.0 will be conducted immediately after the completion of the intervention, and at 1-, 3- and 6-month follow-up via telephone interview.
  The PedsQL 4.0 will be used to assess participants' QoL. This scale includes 23 items that can be categorised into four subscales, including physical functioning, emotional functioning, social functioning, and school functioning. Participants will asked to rate their experience in the past 1 month using a 5-point scale. All items will be reverse scored and linearly transformed into a 0- to 100-point scale. Higher scores represent better quality of life. This scale has been extensively applied in studies among paediatric oncology populations and has well-established psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, phd, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University,, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided